CLINICAL TRIAL: NCT02516150
Title: Effect of Ethanol Intoxication on the Anti-hypoglycemic Action of Glucagon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001323
Record Dates: First submitted 2015-07-28; First posted 2015-08-05 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; Bionic Pancreas; Artificial Pancreas; Insulin; Glucagon; Alcohol; Alcohol Clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Ethanol; Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glucagon with Ethanol (Experimental): Volunteers will receive an infusion of IV ethanol that will increase their BAC (blood alcohol content) to 0.1. Once their BAC has stabilized at 0.1%, 50 micrograms of glucagon will be administered via subcutaneous injection.
  Interventions: Drug: Ethanol; Drug: Glucagon
- Glucagon without Ethanol (Active Comparator): Volunteers will not receive an infusion of IV ethanol at this visit. 50 micrograms of glucagon will be administered via subcutaneous injection.
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Ethanol — IV infusion of ethanol to stabilize BAC (blood alcohol content) at 0.1%
  Other Names: Ethyl Alcohol; Alcohol
  Arms: Glucagon with Ethanol
Drug: Glucagon — injection of 50 micrograms of glucagon

SUMMARY:
This study will test the hypothesis that a BAC (blood alcohol content) of 0.1% will not significantly alter the anti-hypoglycemic effect of mico-dose glucagon in individuals with type 1 diabetes.

DETAILED DESCRIPTION:
This study will test the hypothesis that a BAC (blood alcohol content) of 0.1% will not significantly alter the anti-hypoglycemic effect of mico-dose glucagon in individuals with type 1 diabetes. The study will aim to quantify the effect of a blood alcohol content on the anti-hypoglycemic efficacy of glucagon using a hyperinsulinemic -normoglycemic clamp technique in volunteers with type 1 diabetes in a randomized crossover trial.

ELIGIBILITY:
* Inclusion Criteria:

  * Age 21 to 80 years old with type 1 diabetes for at least one year.
  * Diabetes managed using an insulin infusion pump using rapid-acting insulin such as insulin aspart (NovoLog), insulin lispro (Humalog), or insulin glulisine (Apidra) for at least one week prior to enrollment.
  * Alcohol exposure on at least one occasion in the last year consisting of at least 4 drinks in one sitting.
* Exclusion Criteria:

  * Unable to provide informed consent.
  * Unable to comply with study procedures.
  * Unable to refrain from the consumption of alcohol at least 24 hours prior to study start.
  * Current participation in another diabetes-related clinical trial that, in the judgment of the principle investigator, will compromise the results of the clamp study or the safety of the subject.
  * Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception.
  * Aldehyde dehydrogenase deficiency as determined by a screening questionnaire
  * End stage renal disease on dialysis (hemodialysis or peritoneal dialysis).
  * History of pheochromocytoma (because glucagon has been reported to precipitate hypertensive crisis in the setting of pheochromocytoma). Fractionated metanephrines will be tested in patients with a history increasing the risk for a catecholamine secreting tumor:
  * Paroxysms of tachycardia, pallor, or headache. Personal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease, Episodic or treatment of refractory (requiring 4 or more medications to achieve normotension) hypertension.
  * History of adverse reaction to glucagon (including allergy) besides nausea, vomiting, or headache.
  * Inadequate venous access as determined by study nurse or physician at time of screening.
  * Liver failure or cirrhosis
  * Hemoglobin < 12 gm/dl.
  * History of problem drinking or alcoholism, regardless of whether active or in remission.
  * Use of benzodiazepines or barbiturates or opiates or other central nervous system depressant drugs that could act synergistically with ethanol to lower the level of consciousness
  * Any other factors that, in the judgment of the principal investigator, would interfere with the safe completion of the study procedures.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Diabetes Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 subjects were enrolled. 8 subjects were ineligible to participate, 1 subject withdrew consent, and 2 subjects were not able to be scheduled to participate. 15 subjects participated in both visits.
Groups:
- All Subjects: All subjects enrolled
Period: Overall Study
Arm/Group | All Subjects
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 1
  Unknown or Not Reported | 1
Diabetes Duration [Mean (Standard Deviation); unit: years] | 28.4 (17.1)

OUTCOME MEASURES:

1. Primary Outcome: AOCGIR (Area Over the Curve for Glucose Infusion Rate)
Description: Area over the curve for the glucose infusion rate in the hour following a subcutaneous glucagon dose with a blood alcohol content of 0 vs 0.1%
Time Frame: 1 Day Visit (approximately 8 to 11 hours)
Measure: Mean (Standard Deviation); unit: mg*minute/dl
Arm/Group | Glucagon With Ethanol | Glucagon Without Ethanol
Number analyzed (Participants) | 15 | 15
mg*minute/dl | 1996 (1259) | 1981 (938)

2. Secondary Outcome: Maximum Change in GIR (Glucose Infusion Rate) From Baseline
Description: This outcome is measuring the maximum change in the glucose infusion rate from the GIR at the time of the injection through the 90 minutes after the glucagon injection in the presence and absence of ethanol. The glucose infusion rate is adjusted up to every two minutes throughout the clamp, and for 90 minutes total after the glucagon injection.
Time Frame: 1 Day Visit (approximately 8 to 11 hours)
Measure: Mean (Standard Deviation); unit: ml/hour
Arm/Group | Glucagon With Ethanol | Glucagon Without Ethanol
Number analyzed (Participants) | 15 | 15
ml/hour | 83.0 (35.2) | 101.7 (38.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected by subject report throughout the duration of each clamp visit, which was up to 12 hours long.
Arm/Group | Glucagon With Ethanol | Glucagon Without Ethanol
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucagon With Ethanol (N=15) | Glucagon Without Ethanol (N=15)
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Subject reported a headache, which they rated 4 on a scale of 0-10
Chest tightness (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blurred vision/dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT02516150/Prot_SAP_000.pdf